CLINICAL TRIAL: NCT00958360
Title: VA Low Vision Intervention Trial (LOVIT) II
Brief Title: Low Vision Intervention Trial II (LOVIT II)
Acronym: LOVIT II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C6958-R
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Central Vision Loss From Macular Diseases
Keywords: vision, low
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Interdisciplinary Low Vision Rehabilitation: Low vision examination, prescription and dispensing of low vision devices, low vision therapy and homework.
  Interventions: Other: Interdisciplinary Low Vision Service
- Arm 2 (Active Comparator): Basic Low Vision Care: Low vision examination, prescription and dispensing of low vision devices without low vision therapy or assigned homework.
  Interventions: Other: Basic Low Vision Service

INTERVENTIONS:
Other: Interdisciplinary Low Vision Service — Services are provided by optometrist(s) and low vision therapist(s), and include low vision therapy to improve use of remaining vision and low vision devices, and structured homework to practice use of low vision devices that are prescribed and dispensed.
  Other Names: Interdisciplinary Low Vision Rehabilitation
  Arms: Arm 1
Other: Basic Low Vision Service — Service is provided by the optometrist alone and includes demonstration of low vision device use and maintenance of prescribed low vision devices, without low vision therapy or homework and with less contact time.
  Other Names: Basic Low Vision Rehabilitation
  Arms: Arm 2

SUMMARY:
This study will determine if the interdisciplinary team low vision rehabilitation program is more effective than basic low vision care provided by an optometrist working alone in improving visual reading ability in veterans with macular diseases and best corrected visual acuity of 20/50 to 20/200.

DETAILED DESCRIPTION:
Key Questions: The purpose of our proposed single-masked multicenter randomized controlled trial is to determine if the Interdisciplinary Team approach to low vision service delivery is more effective than the Basic Low Vision Service in improving visual reading ability for 330 veterans with macular diseases and best corrected visual acuity of 20/50-20/200. Effectiveness will be measured with the Veterans Affairs Low Vision Visual Functioning Questionnaire (VA LV VFQ-48), a valid and reliable questionnaire that is administered by telephone to capture changes in patients' self-report of their difficulty reading and performing other daily living activities affected by visual impairment before and after rehabilitation. The primary outcome measure is the comparison of changes in patients' visual reading ability on the VA LV VFQ-48 after they receive low vision care from the Interdisciplinary Team or Basic Low Vision Care program. The secondary outcome measures are comparisons of changes in other VA LV VFQ-48 visual ability scores (overall, mobility, visual information processing, visual motor skills). Hypothesis: The improvement in visual reading ability measured with the VA LV VFQ-48 will be larger for patients who received low vision services from the Interdisciplinary Team than for patients who received the Basic Low Vision Service. Specific Aims:(1) Compare the mean changes in patients' visual reading ability (estimated from patients' difficulty ratings of reading items on the VA LV VFQ-48 before and after low vision service delivery) in the Interdisciplinary Team and Basic Low Vision Care Programs.(2) Compare the mean changes in visual ability [patients' difficulty ratings of other items on the VA LV VFQ-48 (mobility, visual information processing, visual motor skills) before and after low vision service delivery] in the Interdisciplinary Team and Basic Low Vision Care programs.(3). Identify the characteristics of patients who benefit from the Interdisciplinary Team and Basic Low Vision Service. (4). Conduct an economic evaluation to compare the costs and cost effectiveness of the Interdisciplinary Team and Basic Low Vision Service.

ELIGIBILITY:
Inclusion Criteria:

* Primary eye diagnosis (better seeing Eye) macular disease
* Best-corrected visual acuity (better seeing eye) 20/50-20/200

Exclusion Criteria:

* Does not have a telephone
* Does not speak English
* Has received interdisciplinary low vision services
* English literacy less that 5th grade reading level
* Failed TICS
* Unable or unwilling to attend required clinic visits
* Severe hearing impairment preventing administration of telephone questionnaires
* Planned cataract extraction in next 4 months
* Visual fields contracted to diameter of 20 degrees in better-seeing eye
* Vitreous hemorrhage or serous hemorrhagic detachment of macula
* CNVM treated with fewer than 3 anti-VEGF injections
* Diabetic macular edema (DME) treated with focal/grid laser within the last two months
* DME treated with intravitreal injections of anti-VEGF or intravitreal triamcinolone acetonide (IVTA) within the last two months
* Cystoid macular edema (CME) treated with topical (non-steroidal anti-inflammatory drugs) NSAIDS, topical steroids or IVTA within the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2010-08; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Stelmack, OD MPH, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (7):
- United States (7):
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Dayton VA Medical Center, Dayton, OH, Dayton, Ohio
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

REFERENCES:
- [Background] Stelmack JA, Tang XC, Reda DJ, Stroupe KT, Rinne S, Massof RW; LOVIT II Study Group. VA LOVIT II: a protocol to compare low vision rehabilitation and basic low vision. Ophthalmic Physiol Opt. 2012 Nov;32(6):461-71. doi: 10.1111/j.1475-1313.2012.00933.x. Epub 2012 Sep 7. PMID 22958237
- [Derived] Stelmack JA, Tang C, Wei Y, Rose K, Ballinger R, Whitman O, Chronister C, Sayers S, Massof RW; LOVIT II Study Group. Veterans Affairs Low-vision Intervention Trial II: One-year Follow-up. Optom Vis Sci. 2019 Oct;96(10):718-725. doi: 10.1097/OPX.0000000000001428. PMID 31592954
- [Derived] Stroupe KT, Stelmack JA, Tang XC, Wei Y, Sayers S, Reda DJ, Kwon E, Massof RW; LOVIT II Study Group. Economic Evaluation of Low-Vision Rehabilitation for Veterans With Macular Diseases in the US Department of Veterans Affairs. JAMA Ophthalmol. 2018 May 1;136(5):524-531. doi: 10.1001/jamaophthalmol.2018.0797. PMID 29800250
- [Derived] Stelmack JA, Tang XC, Wei Y, Wilcox DT, Morand T, Brahm K, Sayers S, Massof RW; LOVIT II Study Group. Outcomes of the Veterans Affairs Low Vision Intervention Trial II (LOVIT II): A Randomized Clinical Trial. JAMA Ophthalmol. 2017 Feb 1;135(2):96-104. doi: 10.1001/jamaophthalmol.2016.4742. PMID 27978569

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2,051 patients were screened, of whom 1,728 were excluded (1,706 ineligible per chart review and 22 ineligible after screening).
Groups:
- Interdisciplinary Low Vision Rehabilitation Group: Interdisciplinary Low Vision Rehabilitation: Low vision examination, prescription and dispensing of low vision devices, low vision therapy and homework.
  Interdisciplinary Low Vision Service: Services are provided by optometrist(s) and low vision therapist(s), and include low vision therapy to improve use of remaining vision and low vision devices, and structured homework to practice use of low vision devices that are prescribed and dispensed.
- Basic Low Vision Care Group: Basic Low Vision Care: Low vision examination, prescription and dispensing of low vision devices without low vision therapy or assigned homework.
  Basic Low Vision Service: Service is provided by the optometrist alone and includes demonstration of low vision device use and maintenance of prescribed low vision devices, without low vision therapy or homework and with less contact time.
Period: Overall Study
Arm/Group | Interdisciplinary Low Vision Rehabilitation Group | Basic Low Vision Care Group
Started | 163 | 160
Completed | 152 | 150
Not Completed | 11 | 10
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Death | 6 | 7
Not completed — Physician Decision | 2 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interdisciplinary Low Vision Rehabilitation Group | Basic Low Vision Care Group | Total
Number analyzed (Participants) | 163 | 160 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.1 (10.8) | 79.2 (10.1) | 79.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 158 | 156 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 157 | 152 | 309
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 6 | 6
  Black or African American | 15 | 10 | 25
  White | 148 | 144 | 292
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Changes in Visual Reading Ability From Baseline to Four Months Later Measured With 48 Item VA Low Vision Visual Functioning Questionnaire
Description: The range of scores for the Visual Reading Ability subscale of the VA Low Vision Visual Functioning Questionnaire is 0 to 3.5 logits (log odds ratio). A higher score indicates better ability or less difficulty performing activities.
Time Frame: changes from baseline to 4 months later
Measure: Mean (Standard Deviation); unit: logits
Arm/Group | Interdisciplinary Low Vision Rehabilitation Group | Basic Low Vision Care Group
Number analyzed (Participants) | 163 | 160
logits | 1.29 (1.66) | 0.95 (1.46)
Statistical Analysis 1: Comparison: Interdisciplinary Low Vision Rehabilitation Group vs Basic Low Vision Care Group; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

2. Secondary Outcome: Comparison of Changes in Mobility From Baseline to Four Months Later Measured With 48 Item VA Low Vision Visual Functioning Questionnaire
Description: The range of scores for the Mobility subscale of the VA Low Vision Visual Functioning Questionnaire is 0 to 3.5 logits (log odds ratio). A higher score indicates better ability or less difficulty performing activities.
Time Frame: changes from baseline to 4 months later
Measure: Mean (Standard Deviation); unit: logits
Arm/Group | Interdisciplinary Low Vision Rehabilitation Group | Basic Low Vision Care Group
Number analyzed (Participants) | 163 | 160
logits | 0.31 (1.15) | 0.12 (1.16)
Statistical Analysis 1: Comparison: Interdisciplinary Low Vision Rehabilitation Group vs Basic Low Vision Care Group; Test type: Superiority or Other; p = 0.13, t-test, 2 sided

3. Secondary Outcome: Comparison of Changes in Visual Information Processing From Baseline to Four Months Later Measured With 48 Item VA Low Vision Visual Functioning Questionnaire
Description: The range of scores for the Visual Information Processing subscale of the VA Low Vision Visual Functioning Questionnaire is 0 to 3.5 logits (log odds ratio). A higher score indicates better ability or less difficulty performing activities.
Time Frame: changes from baseline to 4 months later
Measure: Mean (Standard Deviation); unit: logits
Arm/Group | Interdisciplinary Low Vision Rehabilitation Group | Basic Low Vision Care Group
Number analyzed (Participants) | 163 | 160
logits | 0.67 (1.21) | 0.40 (1.13)
Statistical Analysis 1: Comparison: Interdisciplinary Low Vision Rehabilitation Group vs Basic Low Vision Care Group; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

4. Secondary Outcome: Comparison of Changes in Visual Motor Skills From Baseline to Four Months Later Measured With 48 Item VA Low Vision Visual Functioning Questionnaire
Description: The range of scores for the Visual Motor Skills subscale of the VA Low Vision Visual Functioning Questionnaire is 0 to 3.5 logits (log odds ratio). A higher score indicates better ability or less difficulty performing activities.
Time Frame: changes from baseline to 4 months later
Measure: Mean (Standard Deviation); unit: logits
Arm/Group | Interdisciplinary Low Vision Rehabilitation Group | Basic Low Vision Care Group
Number analyzed (Participants) | 163 | 160
logits | 0.77 (1.47) | 0.40 (1.19)
Statistical Analysis 1: Comparison: Interdisciplinary Low Vision Rehabilitation Group vs Basic Low Vision Care Group; Test type: Superiority or Other; p = 0.013, t-test, 2 sided

5. Secondary Outcome: Comparison of Overall Visual Ability From Baseline to Four Months Later Measured With 48 Item VA Low Vision Visual Functioning Questionnaire
Description: The range of scores for the Overall Visual Ability subscale of the VA Low Vision Visual Functioning Questionnaire is 0 to 3.5 logits (log odds ratio). A higher score indicates better ability or less difficulty performing activities.
Time Frame: changes from baseline to 4 months later
Measure: Mean (Standard Deviation); unit: logits
Arm/Group | Interdisciplinary Low Vision Rehabilitation Group | Basic Low Vision Care Group
Number analyzed (Participants) | 163 | 160
logits | 0.70 (1.06) | 0.43 (0.89)
Statistical Analysis 1: Comparison: Interdisciplinary Low Vision Rehabilitation Group vs Basic Low Vision Care Group; Test type: Superiority or Other; p = 0.013, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from inception of the study to 4-month follow-up.
Description: This is a low risk non-interventional study. Adverse events were pre-specified in the case report forms and assessed at the 4-month follow-up interview by self-reporting by participants or notification by a family member.
Arm/Group | Interdisciplinary Low Vision Rehabilitation Group | Basic Low Vision Care Group
Serious Adverse Events (participants affected / at risk) | 27/163 | 29/160
Other Adverse Events (participants affected / at risk) | 10/163 | 1/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interdisciplinary Low Vision Rehabilitation Group (N=163) | Basic Low Vision Care Group (N=160)
Non-study related Death (General disorders) | 7 | 8
Non-study related Prolonged Hospitalization (Cardiac disorders) | 4 | 2
Non-study related Prolonged Hospitalization (Endocrine disorders) | 0 | 1
Non-study related Prolonged Hospitalization (Eye disorders) | 0 | 1
Non-study related Prolonged Hospitalization (Gastrointestinal disorders) | 2 | 1
Non-study related Prolonged Hospitalization (General disorders) | 5 | 9
Non-study related Prolonged Hospitalization (Injury, poisoning and procedural complications) | 1 | 3
Non-study related Prolonged Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-study related Prolonged Hospitalization (Renal and urinary disorders) | 2 | 0
Non-study related Prolonged Hospitalization (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Non-study related Prolonged Hospitalization (Vascular disorders) | 3 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interdisciplinary Low Vision Rehabilitation Group (N=163) | Basic Low Vision Care Group (N=160)
eye hemorrhage (Eye disorders) | 3 | 0
CME (Eye disorders) | 7 | 0
other health reason (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes